CLINICAL TRIAL: NCT06265285
Title: Pilot Single-Arm, Pragmatic Trial of In-Home Versus In-Clinic Subcutaneous Nivolumab Administration Through Cancer CARE (Connected Access and Remote Expertise) Beyond Walls (CCBW) Program
Brief Title: Comparison of In-Home Versus In-Clinic Administration of Subcutaneous Nivolumab Through Cancer CARE (Connected Access and Remote Expertise) Beyond Walls (CCBW) Program
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC230716; NCI-2024-00637 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-009663 (Other: Mayo Clinic Institutional Review Board); MC230716 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2024-02-02; First posted 2024-02-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Advanced Esophageal Squamous Cell Carcinoma; Advanced Renal Cell Carcinoma; Clinical Stage II Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IIB Cutaneous Melanoma AJCC v8; Clinical Stage IIC Cutaneous Melanoma AJCC v8; Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage III Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Clinical Stage IV Esophageal Squamous Cell Carcinoma AJCC v8; Esophageal Carcinoma; Gastroesophageal Junction Adenocarcinoma; Hepatocellular Carcinoma; Locally Advanced Urothelial Carcinoma; Lung Non-Small Cell Carcinoma; Malignant Solid Neoplasm; Metastatic Colorectal Carcinoma; Metastatic Cutaneous Melanoma; Metastatic Esophageal Squamous Cell Carcinoma; Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Urothelial Carcinoma; Recurrent Esophageal Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Unresectable Cutaneous Melanoma; Unresectable Esophageal Squamous Cell Carcinoma; Urothelial Carcinoma; Unresectable Urothelial Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Melanoma; Esophageal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Transitional Cell; Carcinoma, Renal Cell | interventions — Home Care Services; House Calls; Nivolumab; Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Health services research (in-clinic and at-home nivolumab) (Experimental): Patients receive nivolumab SC on day 1 of each cycle. Cycles repeat every 28 days in clinic for 2 cycles, then at home by a HHNP for 4 cycles, followed by either in-clinic or at-home administration for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients receive in-home visits by a home health nurse and undergo remote patient monitoring including vital sign measurements and condition-specific symptom assessments throughout the study.
  Interventions: Other: Home Health Encounter; Biological: Nivolumab; Procedure: Patient Monitoring; Other: Questionnaire Administration

INTERVENTIONS:
Other: Home Health Encounter — Receive in-home visits by a home health nurse
  Other Names: HH; Home; Home Care Visit; Home Health
Biological: Nivolumab — Given SC
  Other Names: ABP 206; BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Procedure: Patient Monitoring — Undergo remote patient monitoring
  Other Names: medical monitoring; monitor
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial compares the impact of subcutaneous (SC) nivolumab given in an in-home setting to an in-clinic setting on cancer care and quality of life. Currently, most drug-related cancer care is conducted in clinic type centers or hospitals which may isolate patients from family, friends and familiar surroundings for many hours per day. This separation adds to the physical, emotional, social, and financial burden for patients and their families. Traveling to and from medical facilities costs time, money, and effort and can be a disadvantage to patients living in rural areas, those with low incomes or poor access to transport. Studies have shown that cancer patients often feel more comfortable and secure being cared for in their own home environments. SC nivolumab in-home treatment may be safe, tolerable and/or effective when compared to in-clinic treatment and may reduce the burden of cancer and improve the quality of life in cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the change in patient-reported rating of Cancer Connected Access and Remote Expertise (CARE) after 8 weeks in clinic compared to the same rating after 8 weeks at home.

SECONDARY OBJECTIVES:

I. Evaluate patient preference for location of cancer treatment administration, in the clinic or in the home.

II. Longitudinally assess patient-reported function and global health/quality of life.

III. Longitudinally assess patient-reported symptoms. IV. Assess the safety of cancer directed therapy when administered at home by a home health provider with remote patient monitoring and command center support.

V. Describe emergency room visits and hospitalizations over the course of the study.

VI. Describe overall survival (data collected out to 1 year).

TERTIARY OBJECTIVE:

I. Assess the cost outcomes related to patient treatment in the clinic or in the home.

OUTLINE:

Patients receive nivolumab SC on day 1 of each cycle. Cycles repeat every 28 days in clinic for 2 cycles, then at home by a home health nursing provider (HHNP) for 4 cycles, followed by either in-clinic or at-home administration for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients receive in-home visits by a home health nurse, undergo remote patient monitoring including vital sign measurements and condition-specific symptom assessments throughout the study.

After completion of study treatment, patients are followed up at days 30 and 100, then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed malignancies for which treatment with intravenous nivolumab is currently Food and Drug Administration (FDA) approved and who are recommended to initiate a new treatment regimen with single agent intravenous (IV) nivolumab by their treating oncologist for any of the indications outlined below and who are willing to switch to subcutaneous nivolumab. Additionally, patients who are currently receiving single-agent IV nivolumab are eligible, provided they transition to subcutaneous nivolumab on-study, with their first subcutaneous (subQ) dose administered on cycle 1, day 1 of the study.

  * Single agent nivolumab administered in the adjuvant setting for one of the following indications:

    * Completely resected stage IIB/C, III or IV melanoma
    * Urothelial carcinoma status post radical resection and have a high risk of recurrence
    * Completely resected esophageal or gastroesophageal junction carcinoma with residual pathologic disease in adult patients who have received neoadjuvant chemoradiotherapy (CRT)
  * Single agent nivolumab for advanced/metastatic cancer for one or more of the following indications:

    * Renal cell carcinoma (RCC) patients who have received prior anti-angiogenic therapy
    * Non-small cell lung cancer (NSCLC) with progression on or after platinum-based chemotherapy (Note: patients with EGFR or ALK genomic tumor aberrations should have disease progression on FDA-approved therapy for these aberrations prior to receiving nivolumab)
    * Unresectable advanced, recurrent or metastatic esophageal squamous cell carcinoma (ESCC) after prior fluoropyrimidine- and platinum-based chemotherapy
    * Unresectable or metastatic cutaneous melanoma
    * Locally advanced or metastatic urothelial carcinoma who have disease progression during or following platinum-containing chemotherapy or have disease progression within 12 months of neoadjuvant or adjuvant treatment with platinum-containing chemotherapy
    * Unresectable or metastatic urothelial carcinoma, as first-line treatment in combination with cisplatin and gemcitabine.

      * Subcutaneous nivolumab to be initiated as monotherapy following six cycles of cisplatin + gemcitabine
    * Recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) with disease progression on or after platinum-based therapy
    * Microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) metastatic colorectal cancer (CRC) that has progressed following treatment with a fluoropyrimidine, oxaliplatin, and irinotecan
  * Patients transitioning to maintenance nivolumab and who are willing to switch to subcutaneous nivolumab after completion of Ipilimumab and nivolumab combination therapy for one or more of the indications listed below (Note: patients who discontinue ipilimumab for immune-related toxicities, but are deemed to be eligible to continue on single agent nivolumab maintenance by their treating oncologist are eligible):

    * First-line treatment of adult patients with intermediate or poor risk advanced renal cell carcinoma (RCC)
    * Unresectable or metastatic cutaneous melanoma
    * Hepatocellular carcinoma (HCC) previously treated with sorafenib
    * Microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) metastatic colorectal cancer (CRC) that has progressed following treatment with a fluoropyrimidine, oxaliplatin, and irinotecan
  * Single agent nivolumab administered in the adjuvant setting following neoadjuvant nivolumab with platinum doublet chemotherapy for patients with resectable (tumors ≥ 4 cm and/or node positive) non-small cell lung cancer (NSCLC) and no known epidermal growth factor receptor (EGFR) mutations or anaplastic lymphoma kinase (ALK) rearrangements
* Patients have recovered from the effects of any previous chemotherapy, immunotherapy, other prior systemic anticancer therapy, radiotherapy, and/or surgery (i.e., residual toxicity no worse than grade 1 [grade 2 treatment-associated peripheral neuropathy, grade 2 fatigue and/or any grade of alopecia are acceptable assuming all other inclusion criteria are met]) before registration
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Aspartate transaminase (AST) values ≤ 3 × the upper limit of normal (ULN). For patients with documented baseline liver metastasis, the following limits will apply: 5 × ULN for transaminase
* Alanine transaminase (ALT) values ≤ 3 x the upper limit of normal (ULN). For patients with documented baseline liver metastasis, the following limits will apply: 5 x ULN for transaminase
* Serum total bilirubin values of ≤ 1.5 x ULN ( ≤ 2 x ULN for patients with known Gilbert's syndrome). For patients with documented baseline liver metastasis, the following limits will apply: 2 x ULN for bilirubin
* Absolute neutrophil count (ANC) of ≥ 1500/μL
* Platelet count of ≥ 100,000/μL
* Hemoglobin of ≥ 9 g/dL (patients may be transfused to this level, if necessary, but transfusion must occur > 1 week prior to registration)
* Serum creatinine ≤ 2.0 x the ULN for the reference laboratory or a calculated creatinine clearance of ≥ 30 mL/min by the Cockcroft-Gault Equation measured ≤ 7 days prior to registration
* Patients are residing ≤ 35 miles of clinic (hub) or within the area serviced by supplier and paramedic network
* Residence has Wi-Fi to enable a reliable connection with the remote command center
* Patients have signed Informed Consent Form (ICF)
* Patients are willing and able to comply with the study protocol in the investigator's judgment
* Patients are able and willing to complete study questionnaire(s) by themselves or with assistance
* Women of childbearing potential (WOCBP) must:

  * Have a negative pregnancy test (serum or urine) ≤ 3 days before the first dose of study drug
  * Be agreeable to use a contraceptive method that is highly effective during the intervention period and for at least 5 months after the last dose and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction for the same time period

Exclusion Criteria:

* Patients receiving any other investigational or standard of care agent which would be considered as a treatment for the primary neoplasm and is not part of the eligible treatment regimen
* Patients requiring 24/7 assistance with activities of daily living (ADLs)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Myocardial infarction ≤ 6 months
  * Wound healing disorder
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Patients with any severe infection ≤ 4 weeks prior to registration including, but not limited to, hospitalization for complications of infections
* Patients with an active, known or suspected autoimmune disease. Patients with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. Patients with vitiligo, Graves' disease, or psoriasis not requiring systemic treatment within the past 30 days are not excluded. Patients with celiac disease controlled with diet modification are not excluded
* Patients with a condition requiring systemic treatment with either corticosteroids ( > 10 mg daily prednisone equivalent) ≤ 14 days or other immunosuppressive medications ≤ 30 days prior to registration. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active ≤ 2 years prior to registration (i.e., participants with a history of prior malignancy are eligible if treatment was completed at least 2 years before randomization/treatment assignment and the patient has no evidence of disease). Participants with history of prior early stage basal/squamous cell skin cancer or non-invasive or in situ cancers that have undergone definitive treatment at any time are also eligible
* Patients have undergone prior solid organ and/or non-autologous hematopoietic stem cell or bone marrow transplant
* Patients with active brain metastases or leptomeningeal metastases, aside from the exceptions below. Participants with brain metastases are eligible if they are:

  * Asymptomatic
  * Have been treated and participants have neurologically returned to baseline (except for residual signs or symptoms related to the central nervous system [CNS] treatment), and
  * There is no MRI evidence of progression for at least 4 weeks after CNS directed therapy is complete and ≤ 28 days prior to registration
  * In addition, participants must have been either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent) for at least 2 weeks prior to registration
* Participants with brain disease treated with whole brain radiation
* Anticipation of the need for major surgery during the course of study treatment
* Participants who are pregnant or breastfeeding
* Treatment with any live attenuated vaccines ≤ 30 days of registration (vaccines that are not live attenuated are allowed, including COVID-19 vaccine)
* Known human deficiency virus (HIV) positive with an AIDS defining opportunistic infection within the last year, or a current CD4 count < 350 cells/uL, aside from the exceptions below. Participants with HIV are eligible if:

  * They have received antiviral therapy (ART) for at least 4 weeks prior to treatment assignment as clinically indicated while enrolled in the study
  * They continue on ART as clinically indicated while enrolled on study
  * CD4 counts and viral load are monitored per standard of care by a local healthcare provider
* History of allergy or hypersensitivity to study drug components
* Any positive test result for hepatitis B virus (HBV) indicating presence of virus (e.g., hepatitis B surface antigen [HBsAg, Australia antigen]) positive
* Any positive test result for hepatitis C virus (HCV) indicating presence of active viral replication (detectable HCV-ribonucleic acid [RNA]). Note: Participants with positive HCV antibody and an undetectable HCV RNA are eligible to enroll

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in patient-reported rating of Cancer CARE Cancer Connected Access and Remote Expertise (CARE) after 8 weeks | At baseline and up to 24 weeks of in clinic or at home care
  Measured using the Consumer Assessment of Healthcare Providers and Systems (CAHPS) Cancer Care Survey assessing "your overall cancer care experience," answered on a scale of 0-10 where 0 is the worst experience possible and 10 is the best experience possible. The change in patient-reported rating of Cancer CARE after 8 weeks of in clinic care to the same rating after 8 weeks of at home care will be compared.

SECONDARY OUTCOMES:
Patient preferred treatment location | Up to 24 weeks
  The proportion of patients who prefer care at home or express no preference will be computed and compared with the proportion of patients who prefer care in the clinic.
Patient level of comfort with receiving injections at home | Up to 24 weeks
  The proportion of patients who express comfort will be tabulated and a proportion greater than 70% will signify acceptance. Likert patient feedback questions and "Was It Worth It" questions will be described using frequencies and relative frequencies by arm. Numeric analog scale questions will be described using means and standard deviations and compared within patients (if applicable) using paired t-tests. Descriptive estimates at 24 weeks (after 8 weeks of in clinic and 16 weeks of at home care) will be generated throughout.
Patient-reported symptoms - PRO-CTCAE | Up to 24 weeks
  Patient-reported symptoms will be measured using the Patient Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE). In this study, PRO-CTCAE items were chosen based on common symptoms experienced across cancer patients and side effects common with nivolumab. A free-text item will also be included for patients to report other symptoms as willing. Adverse events (AEs) will be tabulated during the 8 weeks in clinic, and during the 8 weeks at home, compared between arms and summarized over the 24 weeks.
Patient-reported function - EORTC QLQ-F17 | Baseline; 8 weeks; 16 weeks; 24 weeks
  Assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Function 17 (EORTC QLQ-F17), a 17-item patient-reported questionnaire about patient ability to function, overall health and quality of life, and perceived financial impact of cancer and its treatment. The first 15 questions are answered on a scale of 1-4 where 1=not at all, 2=a little, 3=quite a bit, and 4=very much. The final two questions (overall health and overall quality of life during the past week) are answered on a 1-7 numeric analogue scale where 1=very poor and 7=excellent.
Patient-reported side effect impact - GP5 | After 8 weeks of in-clinic and 8 weeks of at home care
  Assessed using the Functional Assessment of Chronic Illness Therapy (FACIT) - Item GP5, "I am bothered by side effects of treatment," which is answered on a scale ranging from 0 (Not at all) to 4 (Very Much). Responses will be computed and compared across patients visits. Mean GP5 scores over time will also be explored.
Incidence of Adverse Events (AEs) | At 8 weeks of in-clinic and 8 weeks at home care
  The maximum grade for each type of AE will be summarized using Common Terminology Criteria for Adverse Events version 5.0. The frequency and percentage of grade 3+ AEs will be reported and compared using McNemar's test.
Emergency room visits and hospitalizations | At 8 weeks of in-clinic and at 8 weeks of at home care
  The proportion of patients with an emergency room visit or hospitalization will be computed and compared using McNemar's test. Proportion of patients with emergency room visits or hospitalizations will also be summarized over the entire study.
Overall survival (OS) | Up to one year post study completion
  OS is defined as the time from study entry to death from any cause. OS will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Roxana S. Dronca, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials